CLINICAL TRIAL: NCT00004220
Title: A Phase I Study of Oxaliplatin in Combination With Gemcitabine
Brief Title: Oxaliplatin and Gemcitabine in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067461; P30CA033572 (NIH); CHNMC-PHI-23; CHNMC-PHL-23; NCI-T99-0003
Record Dates: First submitted 2000-01-28; First posted 2003-04-21 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine; Oxaliplatin

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of oxaliplatin and gemcitabine in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose limiting toxicities of gemcitabine in combination with oxaliplatin in patients with advanced malignancies. II. Determine the pharmacokinetics of oxaliplatin and gemcitabine in these patients.

OUTLINE: This is a multicenter, dose escalation study of gemcitabine. Patients receive oxaliplatin IV over 2 hours on day 1 and gemcitabine IV over 30 minutes on days 1 and 8. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of gemcitabine in combination with a fixed dose of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicity.

PROJECTED ACCRUAL: A total of 24-36 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic or unresectable malignancy for which standard therapy does not exist or is no longer effective No greater than 3 prior treatment regimens No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 2 months Hematopoietic: WBC at least 3000/mm3 Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal SGOT/SGPT no greater than 2.5 times upper limit of normal Renal: Creatinine normal OR Creatinine clearance at least 60 mL/min Cardiovascular: No symptomatic congestive heart failure No unstable angina pectoris No cardiac arrhythmia Other: No clinically significant neuropathy Not pregnant or nursing Fertile patients must use effective contraception No allergy to platinum compounds or antiemetics No uncontrolled active infection or other illness

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics No prior radiotherapy to at least 30% of bone marrow At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics Other: No other concurrent investigational agents No other concurrent anticancer therapy No HIV positive patients receiving antiretroviral therapy (HAART)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I. Shibata, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California